CLINICAL TRIAL: NCT03585894
Title: The Role of Inflammation and Vasodilatation in PACAP38-induced Headache Using MRI on Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Hashmat Ghanizada, Principal investigator, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: H-18008313
Record Dates: First submitted 2018-06-28; First posted 2018-07-13 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Sumatriptan; Ketorolac

STUDY DESIGN:
Intervention Model Description: Each participant will receive PACAP28 intravenous infusion over 20 min in both experiment days but treated in randomized order with sumatriptan or ketorolac.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sumatriptan (Other): Sumatriptan 4 mg/mL I.V will be administrated over 10 min
  Interventions: Other: Sumatriptan
- Ketorolac (Active Comparator): Ketorolac 30 mg/mL I.V will be administrated over 10 min
  Interventions: Other: Ketorolac

INTERVENTIONS:
Other: Sumatriptan — Receive intravenous infusion of sumatriptan
  Arms: Sumatriptan
Other: Ketorolac — Receive intravenous infusion of ketorolac
  Arms: Ketorolac

SUMMARY:
Studying Pituitary adenylate cyclase-activating peptide 38 (PACAP38) induced headache effects on extra- and intracerebral arteries and pre-posttreated by sumatriptan and ketorolac assessed by magnetic resonance imaging (MRI) on healthy volunteers.

DETAILED DESCRIPTION:
The purpose of this research project is to investigate the importance of blood vessel (vasodilatation), vessel wall inflammation and blood flow in arteries of headaches triggered by PACAP38 and for headache treated with sumatriptan (migraine medicine) and ketorolac (NSAID). In addition, we will investigate headache-related changes in the brain's network connectivity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Aged 18-50
* 50-100 kg

Exclusion Criteria:

* Tension type headache more than 5 dag /month
* Other primary headaches
* Daily medication except contraceptives
* Drug taken within 4 times the half-life for the specific drug except contraceptives
* Pregnant or lactating women
* Exposure to radiation within the last year
* Headache within the last 24 hours before start of trial
* Hypertension
* Hypotension
* Respiratory or cardiac disease
* Primary relatives with current or previous migraine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Intra-extra cerebral arteries vasodilatation | 120 minutes
  PACAP38 vasodilatation reverse by sumatriptan but not ketorolac. A single-slab 3D time-of-flight (3D TOF) MRA of extra- and intracranial arteries will be acquired as described in previous studies (Amin et al., 2013, 2014). MRA data will be analyzed by LKEB-MRA vessel wall analysis software program. We will measure the circumference of vessels in millimeter in 4 predefined time points (0, 20, 60 and 110 min)
Headache score | 6 hours
  Visual analog Scale

SECONDARY OUTCOMES:
Blood pressure | 2 hours
  vital parameters recorded at hospital phase
Headache characteristics | 24 hours
  Standard headache questionnaire will be used to record headache localization, nausea, photo and phonophobia.
Heart rate | 2 hours
  vital parameters recorded at hospital phase

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

REFERENCES:
- [Derived] Ghanizada H, Al-Karagholi MA, Arngrim N, Morch-Rasmussen M, Metcalf-Clausen M, Larsson HBW, Amin FM, Ashina M. Investigation of sumatriptan and ketorolac trometamol in the human experimental model of headache. J Headache Pain. 2020 Feb 24;21(1):19. doi: 10.1186/s10194-020-01089-3. PMID 32093617